CLINICAL TRIAL: NCT06482229
Title: Postoperative Analgesic Efficacy of Intraperitoneal Bupivacaine, Bupivacaine and Dexmedetomidine With Modified-Pericondrial Approach Thoracoabdominal Nerve Block (M-TAPA) in Laparoscopic Cholecystectomy Surgeries
Brief Title: M-TAPA vs Intraperitoneal Bupivacain vs Intraperitoneal Bupivacain +Dexmedetomidin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sivas State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Balcı, Specialist/Department of Anaesthesiology and Reanimation, Sivas State Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: m-tapa vs intraperiton
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- m-tapa (Experimental)
  Interventions: Procedure: application for postoperative analgesia
- intraperitoneal bupivacain (Experimental)
  Interventions: Procedure: application for postoperative analgesia
- intraperitoneal bupivacain+dexmedetomidin (Experimental)
  Interventions: Procedure: application for postoperative analgesia

INTERVENTIONS:
Procedure: application for postoperative analgesia — three different methods will be applied to reduce patients' postoperative pain

SUMMARY:
Laparoscopic cholecystectomy is a common abdominal surgery in Western countries, favored for its minimal invasiveness, leading to less pain, smaller scars, and quicker recovery. Despite its benefits, it is contraindicated in cases of bleeding disorders, peritonitis, hemodynamic instability, severe heart failure, and advanced COPD. Effective postoperative pain management is crucial for faster recovery, shorter hospital stays, and lower costs, using techniques such as intravenous or intramuscular analgesics, epidural analgesia, and local anesthetic injections like TAP block or M-TAPA block. The TAPA block, introduced in 2019, involves applying local anesthetic to the costochondral junction, affecting thoracoabdominal nerves, with a modified version (M- TAPA) applying anesthetic to the lower surface only. Studies have shown M-TAPA's efficacy in reducing pain and analgesic use postoperatively. Postoperative pain from laparoscopic cholecystectomy mainly arises from inflammation in the gallbladder bed and pneumoperitoneum. This study aims to evaluate the postoperative analgesic efficacy of intraperitoneal bupivacaine, bupivacaine with dexmedetomidine, and M-TAPA block by assessing pain scores and analgesic consumption in a prospective, randomized, double- blind trial with 45 patients. Patients will be assigned to three groups: M- TAPA block, intraperitoneal bupivacaine, and intraperitoneal bupivacaine with dexmedetomidine, with an experienced anesthetist administering the blocks and evaluating outcomes to compare these pain management techniques.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy surgery planned
* ASA #-II-III classification
* Willingness to participate in the study

Exclusion Criteria:

* Bleeding disorders
* Signs of infection at the block application site
* Conversion to open surgery
* Allergy to local anesthetics
* Unstable hemodynamics
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
pain scores | Time Frame: 24 hours after the procedure
  zero meaning "no pain" and 10 meaning "the worst pain imaginable

SECONDARY OUTCOMES:
total analgesic consumption | 24 hours after the procedure
  total rescue analgesic consumption of patients will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Balci, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No